CLINICAL TRIAL: NCT02137148
Title: Observational Study of the Sonic Window Handheld Ultrasound System for Assistance With Vascular Access and Needle Placement
Brief Title: Sonic Window Study Evaluation Plan
Status: Withdrawn | Type: Observational
Why Stopped: Study was cancelled
Sponsor: Analogic Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E-14-542
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Non-palpable Veins
Keywords: Vascular Access; Sonic Window; Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Use of Ultrasound to assist in needle placement — Use of the Sonic Window handheld Ultrasound device to assist in needle placement by providing a coronal image of the patient anatomy.
  Other Names: Sonic Window; SW1000

SUMMARY:
The goals of this study are as follows; evaluation of the products' readiness to market, ascertain initial reactions by target users, evaluate actual use in potential clinical settings and any difficulties encountered with product use and actual venous cannulation.

DETAILED DESCRIPTION:
This study was cancelled

ELIGIBILITY:
Inclusion Criteria:

* Patient Requires needle placement

Exclusion Criteria:

* Under 18 years of age
* Needle placement not required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 adults who require vascular access
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
First Stick Success | 10 minutes
  With this study we want to confirm that The Sonic Window aids in locating and accessing non-palpable veins in a group of up to 50 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Arveh Shander, M.D., Principal Investigator — EHMC
Locations (1):
- Englewood Hospital & Medical Center, Englewood, New Jersey, United States